CLINICAL TRIAL: NCT04446455
Title: A Pilot to Evaluate the Feasibility and Efficacy of a Multifaceted Rehabilitation Intervention
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan F. Bean, Director, New England Geriatric Research Education and Clinical Center, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3014
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Mobility Limitation
Keywords: Rehabilitation; Aging; Mobility Skills; Cognitive Training
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Randomized Pilot Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Power + Cognitive Training (Experimental): Training sessions began with approximately 30 minutes of cognitive training using a desktop computer followed by 40 minutes of functional power training.
  Interventions: Other: InVEST: Increased Velocity Exercise Specific to Task; Other: TAPAT: Tonic and Phasic Alertness Training
- Functional Power Training (Active Comparator): Training sessions began with 40 minutes of functional power training.
  Interventions: Other: InVEST: Increased Velocity Exercise Specific to Task

INTERVENTIONS:
Other: InVEST: Increased Velocity Exercise Specific to Task — Functional Power Training
Other: TAPAT: Tonic and Phasic Alertness Training — Computerized cognitive training.
  Arms: Functional Power + Cognitive Training

SUMMARY:
The goal of this study is to evaluate the efficacy of multifaceted rehabilitation program in Veterans 65 years and older. This study will also examine the neuromuscular and cognitive attributes that contribute to clinically meaningful improvements in mobility; and determine whether a novel mode of cognitive training can enhance cognition among mobility limited primary care Veterans 65 years and older.

DETAILED DESCRIPTION:
This study is a randomized control pilot study. All participants will receive rehabilitative exercise addressing mobility skills. In addition, one group will be will receive additional cognitive training. Randomization is stratified according to screening mobility and cognitive score.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-90
* History of fall in the past year OR difficulty or task modification with climbing one flight of stairs or walking ½ mile (6 blocks)
* Community Dwelling
* Ability to speak and understand English

Exclusion Criteria:

* Presence of a terminal disease (e.g. receiving hospice services, metastatic cancer
* Major medical problem interfering with safe and successful testing (i.e. history of hip replacement with recurrent dislocation; uncontrolled hypertension, use of supplemental oxygen
* Myocardial infarction or major surgery in previous 3 months
* Planned major surgery (e.g. joint replacement)
* Baseline Short Physical Performance Battery Score <4 or >10
* Modified Mini Mental Status Examination score of ≤77 out of 100
* Inability to safely complete the 400 meter walk test

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Late-Life Function and Disability Instrument at 6 weeks | Baseline, 6 weeks
  Function domain and the advanced and basic lower extremity function sub-domains of the Late-Life Function and Disability Instrument

SECONDARY OUTCOMES:
Change from Baseline Figure-of-8 Performance 6 weeks | Baseline, 6 weeks
Change from Baseline 400 Meter Walk Test at 6 weeks | Baseline, 6 weeks
Change from Baseline Short Physical Performance Battery (SPPB) at 6 weeks | Baseline, 6 weeks
  Range: 0-12; higher score better physical performance
Change from Baseline Cognitive Performance at 6 weeks | Baseline, 6 weeks
Change from Baseline Trail Making Test at 6 weeks | Baseline, 6 weeks
Change from Baseline Clock-in-the-Box Test at 6 weeks | Baseline, 6 weeks
Change from Baseline Letter Fluency Test at 6 weeks | Baseline, 6 weeks
Change from Baseline Hopkins Verbal Learning Test at 6 weeks | Baseline, 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No